CLINICAL TRIAL: NCT01202877
Title: A Combination of PKC412 and 5-Azacytidine for the Treatment of Patients With Refractory or Relapsed Acute Leukemia and Myelodysplastic Syndrome (MDS)
Brief Title: PKC412 and 5-Azacytidine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0374; NCI-2012-01896 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2015-07

CONDITIONS: Leukemia
Keywords: Myelodysplastic Syndrome; MDS; Refractory acute leukemias; Relapsed acute leukemia; Acute myeloid leukemia; AML; 5-Azacytidine; Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; PKC412
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-azacytidine + PKC412 (Experimental): 5-azacytidine 75 mg/m2/d subcutaneously (SQ) or by vein (IV) on days 1-7 of a 28 day cycle. PKC412 50 mg by mouth twice daily for 14 days (days 8-21), of every 28 day cycle. Starting with cycle 2, PKC412 administered continuously (daily).
  Interventions: Drug: 5-azacytidine; Drug: PKC412

INTERVENTIONS:
Drug: 5-azacytidine — Starting dose: 75 mg/m2/d subcutaneously (SQ) or by vein (IV) on days 1-7 of a 28 day cycle.
  Other Names: Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
Drug: PKC412 — Starting dose: 50 mg by mouth twice daily for 14 days (days 8-21), of every 28 day cycle. Starting with cycle 2, PKC412 administered continuously (daily).
  Other Names: Midostaurin

SUMMARY:
The goal of this clinical research study is to learn if the combination of PKC412 (also called Midostaurin) and 5-azacytidine can help to control refractory or relapsed acute leukemia and MDS. The safety and best dose of the combination of the drugs will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

PKC412 is designed to block certain receptors (FLT3-Kinase) on cancer cells that are responsible for cancer growth. This may cause the cancer cells to die.

5-azacytidine is designed to cause changes to certain genes that are thought to participate in causing leukemia. These changes are thought to silence these genes so they cannot contribute any longer to sustain the growth of leukemia and MDS.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a part of the study based on when you join.

* If you are one of the first 6 participants, you will receive a pre-planned dose of the study drugs. If 2 participants experience severe side effects, the rest of this group will receive a lower dose.
* If you are not one of the first 6 participants, and fewer than 2 patients had severe side effects in the first group, you will receive the drugs at a higher dose than the first 6 participants.

Study Drug Administration:

You will receive 5-azacytidine by vein over about 30 minutes or through a needle under your skin on Days 1-7 of each 28-day study cycle. Your doctor will decide if you will get the drug by vein or under the skin. You will be required to return to MD Anderson for the first 7 days of every cycle to receive 5-azacytidine.

On Days 8-21 of cycle 1, you will take PKC412 capsules by mouth 2 times a day. Starting with Cycle 2, you will take PKC412 capsules by mouth every day. The research staff will tell you how to take the study drug and you will also be given instructions.

If you have severe side effects from the study drug, the study doctor may decide to stop drug dosing until your side effects improve.

Study Visits:

At every visit, you will be asked about any side effects you have experienced and to list any drugs you may be taking.

* At the start of Cycles 1-2 (+/- 4 days) and then every 2-3 cycles, you will have a complete physical exam.
* Every week during Cycles 1-3 (+/- 4 days) and then every 2-4 weeks, blood (about 1 tablespoon) will be drawn for routine tests and to test your kidney and liver function.
* On Day 28 of Cycle 1 (+/- 4 days) and then every 1-3 cycles, you will have a bone marrow aspirate to check the status of the disease.
* On Day 8 (+/- 1 day) of each cycle for the first cycle before initiation of Midostaurin, then before the start of Midostaurin on Cycle 2, then on Day 1 every 2-3 Cycles, you will have an ECG.
* On Days 8, 15, and 21 of Cycle 1 and Day 1 of Cycle 2, blood (about 1 teaspoon) will be drawn for Pharmacokinetic (PK) testing before you take the study drug.

If you stay on study for longer than 6 months, your doctor will decide what tests and procedures you will have and when they will be performed. At least every 6-12 months you will have a bone marrow aspirate.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

This is an investigational study. PKC412 is not FDA approved or commercially available. It is currently being used for research purposes only. 5-azacytidine is FDA approved and commercially available for the treatment of patients with MDS. The combination of these drugs to treat refractory or relapsed acute leukemia and MDS is investigational.

Up to 54 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS, chronic myelomonocytic leukemia (CMML), AML or biphenotypic or bilineage leukemia who have failed prior therapy. Patients with MDS or CMML should have failed prior therapy with a hypomethylating agent and/or with lenalidomide. Patients with AML should have failed any prior induction therapy or have relapsed after prior therapy, or be previously untreated and unable or unwilling to receive conventional chemotherapy (e.g., patients age >/=65 years). Patients with MDS or CMML who received therapy with a hypomethylating agent and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for AML. The World Health Organization (WHO) classification will be used for AML. Patients with MDS, CMML or AML who have received no prior therapy are eligible if not candidates to receive or refuse standard therapy.
2. Patients must have evidence of FLT3 activating mutations.
3. Age >/= 18 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Status </= 2
5. Adequate liver (bilirubin </= 2x ULN, alanine aminotransferase (ALT) </= 2.5x ULN) and renal (creatinine </= 2x ULN) function
6. Patients must provide written informed consent.
7. Patients must have been off chemotherapy for 2 weeks prior to entering this study, unless there is evidence of rapidly progressive disease, and must have recovered from the toxic effects of that therapy to at least grade 1. Use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy.
8. Women of childbearing potential must practice contraception. Women considered not of childbearing potential include any of the following: no menses for at least 5 years or menses within 5 years but amenorrheic for at least 2 months and luteinizing hormone (LH) and follicular stimulating hormone (FSH) values within normal range (according to definition of postmenopausal for laboratory used) or bilateral oophorectomy or radiation castration and amenorrheic for at least 3 months. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation.
9. **continued from above: Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study.
10. Sexually active males should use a condom during intercourse while taking drug and for 3 months after stopping midostaurin medication. They should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid .
11. Negative urine or serum pregnancy test within 2 weeks.

Exclusion Criteria:

1. Patients with known allergy or hypersensitivity to PKC412, mannitol or 5-azacytidine, or any of their components.
2. Patients who have received any treatment of midostaurin prior to study entry.
3. Patients with known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PKC412.
4. Patients who demonstrated primary resistance to any FLT3 inhibitor or who relapsed while on therapy with a FLT3 inhibitor.
5. Patients with any other known disease (except carcinoma in-situ) concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes with fasting glucose > 200 mg/dl despite optimal management, cardiovascular disease including congestive heart failure (NYHA Class III or IV), myocardial infarction within 6 months and poorly controlled hypertension with systolic > 160 mmHg and diastolic > 100 mmHg, chronic renal disease, or active uncontrolled systemic infection) which could compromise participation in the study.
6. Patients with a known confirmed diagnosis of HIV infection or active viral hepatitis. HIV patients not on specific antiretroviral therapy are eligible for participation.
7. Patients who have had any major surgical procedure within 14 days of Day 1.
8. Patients unwilling or unable to comply with the protocol.
9. Patients with known advanced malignant disease of the central nervous system.
10. Impaired cardiac function including any of the following: Screening ECG with a corrected QT interval (QTc) > 470 msec; Patients with congenital long QT syndrome; History or presence of sustained ventricular tachycardia; Any history of ventricular fibrillation or torsades de pointes; Bradycardia defined as Heart Rate (HR) < 50 bpm; Right bundle branch block + left anterior hemiblock (bifascicular block); Patients with myocardial infarction or unstable angina < 6 months prior to starting study drug; congestive heart failure (CHF) NY Heart Association class III or IV; Patients with an ejection fraction < 50% assessed by multigated radionuclide angiography (MUGA) or echocardiogram (ECHO) scan within 14 days of Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 2, 2011 to October 01, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: There were 57 participants for enrollment, one participant was a screen failure and two withdrew consent without receiving the study drug treatment and are therefore excluded from the study.
Groups:
- Phase I: 5-azacytidine + PKC412 25 mg: 5-azacytidine 75 mg/m2/day subcutaneously (SQ) or by vein (IV) on days 1-7 of a 28 day cycle. PKC412 25 mg orally twice daily for 14 days (days 8-21), of every 28 day cycle. Starting with cycle 2, PKC412 administered continuously (daily).
- Phase I: 5-azacytidine + PKC412 50 mg: 5-azacytidine 75 mg/m2/day subcutaneously (SQ) or by vein (IV) on days 1-7 of a 28 day cycle. PKC412 50 mg orally twice daily for 14 days (days 8-21), of every 28 day cycle. Starting with cycle 2, PKC412 administered continuously (daily).
- Phase II: 5-azacytidine + PKC412: AZA 75 mg/m^2 on days 1-7 and Midostaurin 50 mg bid orally on day 8-21 during the first cycle and continuously thereafter.
Period: Overall Study
Arm/Group | Phase I: 5-azacytidine + PKC412 25 mg | Phase I: 5-azacytidine + PKC412 50 mg | Phase II: 5-azacytidine + PKC412
Started | 6 | 8 | 40
Completed | 6 | 7 | 34
Not Completed | 0 | 1 | 6
Not completed — Disease Progression | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: 5-azacytidine + PKC412 25 mg: 5-azacytidine (AZA) 75 mg/m^2/day subcutaneously (SQ) or by vein (IV) on days 1-7 of a 28 day cycle. PKC412 25 mg orally twice daily for 14 days (days 8-21), of every 28 day cycle. Starting with cycle 2, PKC412 administered continuously (daily).
- Phase I: 5-azacytidine + PKC412 50 mg: AZA 75 mg/m^2/day SQ or IV on days 1-7 of a 28 day cycle. PKC412 50 mg orally twice daily for 14 days (days 8-21), of every 28 day cycle. Starting with cycle 2, PKC412 administered continuously (daily).
- Total: Total of all reporting groups
Arm/Group | Phase I: 5-azacytidine + PKC412 25 mg | Phase I: 5-azacytidine + PKC412 50 mg | Phase II: 5-azacytidine + PKC412 | Total
Number analyzed (Participants) | 6 | 8 | 40 | 54
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 68] | 62 [38 to 85] | 67 [21 to 83] | 65 [21 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 16 | 22
  Male | 4 | 4 | 24 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 40 | 54

OUTCOME MEASURES:

1. Primary Outcome: Participant Best Response Assessed Using Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
Description: Criteria for response per international working group for Myelodysplastic Syndrome (MDS) & acute myeloid leukemia (AML) where responders obtained a complete remission (CR), a CR with incomplete bone marrow recovery (CRi), a morphologic leukemia-free status (MLFS), or a partial remission (PR). CR: <5% bone marrow blasts, neutrophil count>1.0 X10⁹/L, & platelet count>100 X10⁹/L. CRi: all CR criteria except residual neutropenia (<1.0 X10⁹/L) or thrombocytopenia (<100 X10⁹/L). MLFS: <5% blasts in bone marrow regardless of neutrophil & platelet count in peripheral blood. PR: all CR criteria, except reduction> 50% in bone marrow blasts, but still >5%. Clinical responses evaluated using RECIST version 1.1 criteria after every two cycles, with confirmation of clinical response at 4 weeks after achieving response.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Phase I: 5-azacytidine + PKC412 25 mg: AZA 75 mg/m^2/day subcutaneously (SQ) or by vein (IV) on days 1-7 of a 28 day cycle. PKC412 25 mg orally twice daily for 14 days (days 8-21), of every 28 day cycle. Starting with cycle 2, PKC412 administered continuously (daily).
- Phase II: 5-azacytidine + PKC412: AZA 75 mg/m^2 on days 1-7 and PKC412 Midostaurin 50 mg bid orally on day 8-21 during the first cycle and continuously thereafter.
Arm/Group | Phase I: 5-azacytidine + PKC412 25 mg | Phase I: 5-azacytidine + PKC412 50 mg | Phase II: 5-azacytidine + PKC412
Number analyzed (Participants) | 6 | 8 | 40
participants
  Complete Remission (CR) | 0 | 0 | 1
  Complete w/Incomplete Bone Marrow Recovery (CRi) | 1 | 1 | 4
  Morphologic Leukemia-Free Status (MLFS) | 0 | 0 | 6
  Partial Remission (PR) | 0 | 0 | 1

2. Primary Outcome: Overall Response (OR) Within 6 Months
Description: Overall response defined as number of participants with response as follows: (OR = CR [complete response (CR) rate] + CRi [complete remission with incomplete count recovery] + PR [partial remission] + HI [hematologic improvement]) within 6 months of treatment initiation. complete remission (CR), a CR with incomplete bone marrow recovery (CRi), a morphologic leukemia-free status (MLFS), or a partial remission (PR). CR: <5% bone marrow blasts, neutrophil count>1.0 X10⁹/L, & platelet count>100 X10⁹/L. CRi: all CR criteria except residual neutropenia (<1.0 X10⁹/L) or thrombocytopenia (<100 X10⁹/L). MLFS: <5% blasts in bone marrow regardless of neutrophil & platelet count in peripheral blood. PR: all CR criteria, except reduction> 50% in bone marrow blasts, but still >5%.
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Phase I: 5-azacytidine + PKC412 25 mg | Phase I: 5-azacytidine + PKC412 50 mg | Phase II: 5-azacytidine + PKC412
Number analyzed (Participants) | 6 | 8 | 40
participants | 1 | 1 | 12

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of the first protocol-specific intervention with each 21 day cycle until 30 days after the last dose of drug, about 6 months.
Arm/Group | Phase I: 5-azacytidine + PKC412 25 mg | Phase I: 5-azacytidine + PKC412 50 mg | Phase II: 5-azacytidine + PKC412
Serious Adverse Events (participants affected / at risk) | 5/6 | 5/8 | 29/40
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 5-azacytidine + PKC412 25 mg (N=6) | Phase I: 5-azacytidine + PKC412 50 mg (N=8) | Phase II: 5-azacytidine + PKC412 (N=40)
Altered Mental Status (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Pain (General) (General disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Renal Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left Ventricular systolic dysfuction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1) | 3 (3) — Progressive Disease
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Hematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac Other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Complication Surgical medical procedure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pain, Bone/Extremity (General disorders) | 0 (0) | 0 (0) | 3 (3)
Infection from catheter (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Neutropenia Fever (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1)
Infection of blood (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 8 (8)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Wound Infection (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 5-azacytidine + PKC412 25 mg (N=6) | Phase I: 5-azacytidine + PKC412 50 mg (N=8) | Phase II: 5-azacytidine + PKC412 (N=40)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 8 (8) | 40 (40)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 8 (8)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (6)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperbilirubinemia (Investigations) | 2 (2) | 0 (0) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Infections (Infections and infestations) | 4 (4) | 6 (6) | 25 (25)
Nausea/vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6) | 19 (19)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 8 (8) | 40 (40) — Abnormal Absolute Neutrophile Count
Electrocardiogram QTc prolongation (Investigations) | 0 (0) | 0 (0) | 5 (5)
Skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 9 (9)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 5 (5)
Thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 5 (5)
Abnormal liver function test (LFT) (Renal and urinary disorders) | 0 (0) | 0 (0) | 6 (6)
Headache (General disorders) | 1 (1) | 2 (2) | 5 (5)
Low Hemoglobin (Investigations) | 6 (6) | 8 (8) | 40 (40)
Mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 14 (14)
Platelet Increased (Investigations) | 6 (6) | 8 (8) | 40 (40)
Prolongation of QT interval (Investigations) | 0 (0) | 0 (0) | 5 (5) — Electrocardiogram QT corrected interval prolonged

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes